CLINICAL TRIAL: NCT02687633
Title: Early Behavioral Intervention to Improve Social Communication Function in Infants With Tuberous Sclerosis Complex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Shafali Jeste, MD, Assistant Professor in Psychiatry and Neurology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-000699
Record Dates: First submitted 2016-02-10; First posted 2016-02-22 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Tuberous Sclerosis Complex
MeSH Terms: conditions — Tuberous Sclerosis | interventions — Activator Appliances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): The Treatment Group begins the JASPER intervention immediately upon enrollment in the study.
  Interventions: Behavioral: JASPER
- Delayed Treatment Group (Active Comparator): The Delayed treatment group receives the same JASPER intervention as the Treatment Group, but after 6 months of receiving services in the community as usual.
  Interventions: Behavioral: JASPER

INTERVENTIONS:
Behavioral: JASPER — JASPER (Joint Attention, Symbolic Play, Engagement, and Regulation) is a treatment approach based on a combination of developmental and behavioral principles developed by Dr. Connie Kasari and Dr. Amanda Gulsrud at UCLA. It targets the foundations of social communication (joint attention, imitation, play) and uses naturalistic strategies to increase the rate and complexity of social communication.
  Other Names: Joint Attention, Symbolic Play and Engagement Regulation

SUMMARY:
The investigators are running an intervention study for young children with Tuberous Sclerosis Complex (TSC). The study will include free play-based behavioral intervention that may improve social and communication skills in children with TSC. Eligible families will have a child in the age range of 12-36 months, with a diagnosis of TSC. A parent must also be available to attend the weekly intervention sessions at UCLA.

The intervention will focus on teaching caregivers skills to improve the social and communication outcomes of their children. The content of the intervention will be individually tailored to the child's developmental level. The intervention involves pre-assessments, an intervention period of daily 60 minute sessions for 10 days, followed by weekly 60 minute sessions for 10 weeks, and post-assessments. The classroom can have up to 3 parent-child dyad and the curriculum focuses on improving social-communication and play skills.

DETAILED DESCRIPTION:
Most children with Tuberous Sclerosis Complex (TSC) suffer from neurodevelopmental disabilities, including intellectual disability (ID) and autism spectrum disorder (ASD). There is a tremendous need for early intervention for all infants with TSC, with a focus on improving non-verbal cognition and social communication skills. However, no studies have investigated whether early intervention can improve social communication skills in infants with TSC. As a result, families of infants with TSC struggle to receive adequate interventions targeting these areas of development.

The investigators propose to enroll 32 infants and toddlers with TSC to study an evidence-based behavioral intervention in infants with TSC, combining the efforts of investigators with expertise in autism intervention, infant development, and TSC. The proposed intervention study adapts a parent-mediated treatment called JASPER (Joint attention, symbolic play, engagement, regulation) that has successfully improved social communication outcomes in toddlers and young children with ASD.

JASPER intervention will last 3 months, and is split into two phases. Phase 1 occurs for the first 2 weeks of intervention, and consists of daily 1 hour intervention sessions (Monday through Friday) for 2 weeks. After Phase 1, Phase two begins, and consists of 60 minute sessions once a week for 10 weeks. Participants will receive behavioral assessments and EEG across 4 assessment time points during this study: At the start of participation in the study, two weeks into participation of the study, 3 months into participation of the study, and 6 months into participation in the study. The behavioral assessments administered throughout these time points will measure social communication skills, overall cognitive functioning, and non-verbal communication. EEG is sensitive to subtle changes in the brain and may be able to capture responses to treatment prior to clinical or behavioral change, and can inform researchers of the brain basis for the behavioral changes found with intervention. The EEG at each time point will be 30-45 minutes in length, and will require the participant to be awake, as they will watch several short videos on a tv screen while recording EEG data.

There are 2 randomized participation groups in this study, Treatment Group 1, and Treatment Group 2. Treatment group 1 will begin JASPER intervention immediately, and thus will complete the first 3 assessment time points while in intervention, and the 4th assessment time point 3 months after intervention ends. Treatment Group 2 will complete the 4 assessment time points while receiving services as usual in the community, and will begin intervention after the 4th assessment time point. Treatment group 1 will participate in this study for a total of 6 months, and treatment group 2 will participate in the study for a total of 9 months, since they will receive services in the community as usual for 6 months before beginning the 3 month intervention. Group assignment is randomized, and each participant has an equal chance of being assigned to either treatment group.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of Tuberous Sclerosis Complex

Exclusion Criteria:

* A mental age less than 6 months. A plan for epilepsy surgery during the study participation period.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2015-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
change from baseline in Joint Engagement (shared engagement in a play routine) at 2 weeks into study participation, according to the parent caregiver interaction assessment. | 2 weeks
  Parent Caregiver Interaction assesses the amount of time the parent and child spend in engaged in the same play routine.
change from baseline in Joint Engagement (shared engagement in a play routine) at 3 months into study participation, according to the parent caregiver interaction assessment. | 3 months
  Parent Caregiver Interaction assesses the amount of time the parent and child spend in engaged in the same play routine.
change from baseline in Joint Engagement (shared engagement in a play routine) at 6 months into study participation, according to the parent caregiver interaction assessment. | 6 months
  Parent Caregiver Interaction assesses the amount of time the parent and child spend in engaged in the same play routine.

SECONDARY OUTCOMES:
Change from baseline in the amount of time spent in a Joint Attention (the coordination of attention between objects and people for the purpose of sharing) state at 2 weeks | 2 weeks
  ESCS (Early Social Communication Scales) Assessment.
Change from baseline in the amount of time spent in a Joint Attention (the coordination of attention between objects and people for the purpose of sharing) state at 3 months | 3 months
  ESCS (Early Social Communication Scales) Assessment.
Change from baseline in the amount of time spent in a Joint Attention (the coordination of attention between objects and people for the purpose of sharing) state at 6 months | 6 months
  ESCS (Early Social Communication Scales) Assessment.
Change from baseline in Symbolic Play (types of play and level of play) at 2 weeks, according to the Structured Play Assessment (SPA) | 2 weeks
  The Structured Play Assessment measures the child's play level, based on distinct sets of toys that target specific developmental markers of play.
Change from baseline in Symbolic Play (types of play and level of play) at 3 months, according to the Structured Play Assessment (SPA) | 3 months
  The Structured Play Assessment measures the child's play level, based on distinct sets of toys that target specific developmental markers of play.
Change from baseline in Symbolic Play (types of play and level of play) at 6 months, according to the Structured Play Assessment (SPA) | 6 months
  The Structured Play Assessment measures the child's play level, based on distinct sets of toys that target specific developmental markers of play.
Change from baseline at 3 months in developmental quotient, as determined by the Mullen Scales of Early Learning | 3 months
  Cognition will be determined by a Developmental Quotient on a traditional cognitive measure, the Mullen Scales of Early Learning
Change from baseline at 6 months in developmental quotient, as determined by the Mullen Scales of Early Learning | 6 months
  Cognition will be determined by a Developmental Quotient on a traditional cognitive measure, the Mullen Scales of Early Learning
Change from baseline at 2 weeks in the amount of Parent use of social communication support strategies | 2 weeks
  Parent use of social communication support strategies as taught by JASPER will be measured by a parent-child interaction assessment.
Change from baseline at 3 months in the amount of Parent use of social communication support strategies | 3 months
  Parent use of social communication support strategies as taught by JASPER will be measured by a parent-child interaction assessment.
Change from baseline at 6 months in the amount of Parent use of social communication support strategies | 6 months
  Parent use of social communication support strategies as taught by JASPER will be measured by a parent-child interaction assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Shafali Jeste, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Insitute, Los Angeles, California, United States